CLINICAL TRIAL: NCT06312865
Title: Clinical and Demographic Characteristics of Intermittent Exotropia in Egyptian Population
Brief Title: Intermittent Exotropia in Egyptian Population
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud F. Rateb, Principal investigator, Assiut University
Other Study IDs: IXTEGYPT
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Exotropia
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients diagnosed with 8 prism diopters or more exodeviation at distant or near fixation, regardless of age or fusion control (including intermittent exotropia, and constant exotropia).
  Interventions: Device: Ophthalmic exam

INTERVENTIONS:
Device: Ophthalmic exam — include best corrected visual acuity and cycloplegic refraction data

SUMMARY:
Strabismus is one of the most frequent ocular problems among developmentally normal children. The prevalence of strabismus varies among different regions, ranging from 0.06% in Japan to 5.65% in China. Exotropia is reported to be the most prevalent type of deviation in many of these studies. About 48-92% of the exotropic patients have intermittent exotropia (IXT). Jenkins reported that the prevalence of exodeviation was higher in countries near the Equator. Its prevalence is also higher in subequatorial Africa, the Middle East, and East Asia (where there is plenty of sunshine) in comparison to the USA and Central Europe. Intermittent exotropia is a disorder of binocular eye movement control, where one eye intermittently turns outward. The outward deviation is greatest and likely occurs at far distances viewing, when the oculomotor convergence effort is weakest, and occurs frequently when the patient is under stress, tired, ill, or in particular test situations. X(T) can also occur at near as convergence insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with 8 prism diopters or more exodeviation at distant or near fixation, regardless of age or fusion control (including exophora, intermittent exotropia, and constant exotropia).

Exclusion Criteria:

* patients with congenital ocular anomalies or ocular mayopathies. Patients with limitation of ocular motility resulting in strabismus, including neurologic or paralytic disorders, previous ocular surgical history, including strabismus and visually affecting surgeries, or any conditions affecting the central visual acuity, including anterior segment abnormality, cataracts, retinal diseases, or blepharoptosis (ocular sensory disorders), were excluded. When a patient was suspected to visit multiple institutions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian population
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The difference in demographic criteria in Egyptian population | 6 months